CLINICAL TRIAL: NCT04133909
Title: A Multi-center, Randomized, Double-blind, Parallel-group, Placebo-controlled Study of Mepolizumab 100 mg SC as add-on Treatment in Participants With COPD Experiencing Frequent Exacerbations and Characterized by Eosinophil Levels (Study 208657)
Brief Title: Mepolizumab as Add-on Treatment IN Participants With COPD Characterized by Frequent Exacerbations and Eosinophil Level
Acronym: MATINEE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 208657
Expanded Access: NCT00244686 (No longer available)
Record Dates: First submitted 2019-10-18; First posted 2019-10-21 (Actual); Results first posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; Mepolizumab; Exacerbations; MATINEE
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — mepolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mepolizumab 100 mg (Experimental): Participants with Chronic Obstructive Pulmonary Disease (COPD) received a 100 milligrams (mg) dose of mepolizumab as a subcutaneous injection every 4 weeks. Participants remained in the study for an assessment period of minimum of 52 weeks and a maximum of 104 weeks.
  Interventions: Biological: Mepolizumab
- Placebo (Experimental): Participants with COPD received matching placebo as a subcutaneous injection every 4 weeks. Participants remained in the study for an assessment period of minimum of 52 weeks and a maximum of 104 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Mepolizumab — Mepolizumab was a sterile liquid formulation. It was administered as a subcutaneous injection (100 milligrams per milliliter [mg/mL]) delivered once every 4 weeks using a pre-filled safety syringe.
  Arms: Mepolizumab 100 mg
Drug: Placebo — Placebo was a 0.9% sodium chloride solution. It was administered as a subcutaneous injection delivered once every 4 weeks using a pre-filled safety syringe.
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, placebo-controlled, double-blind, parallel group study designed to confirm the benefits of mepolizumab treatment on moderate or severe exacerbations in chronic obstructive pulmonary disease (COPD) participants given as an add on to their optimized maintenance COPD therapy. The maximum duration of participant participation is approximately 109 weeks, consisting of 2 screening visits (up to 3 weeks), a run-in period (up to 2 weeks), and an intervention period of at least 52 weeks and up to 104 weeks. 800 participants will be randomized in a 1:1 ratio to receive mepolizumab 100 milligrams (mg) or placebo every 4 weeks for at least 13 doses (52 weeks treatment period) up to a maximum of 26 doses (104 weeks treatment period). The number of randomized participants may increase up to approximately 1400.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 40 years of age at Screening Visit 1.
* Participants with a peripheral blood eosinophil count of >=300 cells per microliter (μL) from the hematology sample collected at Screening Visit 0 AND a documented historical blood eosinophil count of >=150 cells per μL in the 12 months prior to Screening Visit 0 that meets the following: It must have been measured between 12 months and 1 month prior to Screening Visit 0, and it must not have been measured within 14 days of a COPD exacerbation. Participants with no documented historical blood eosinophil count of >=150 cells per µL must meet this threshold at the Screening Visit 1 assessment.
* Participants with a clinically documented history of COPD for at least 1 year in accordance with the definition by the American Thoracic Society or European Respiratory Society.
* Participants must present with a measured pre- and post-salbutamol Forced expiratory volume in one second (FEV1)/Forced vital capacity (FVC) ratio of <0.70 at Screening Visit 1 to confirm the diagnosis of COPD and with a measured post-salbutamol FEV1>20% and <=80% of predicted normal values calculated using NHANES III reference equations at Screening Visit 1.
* Participants must have a well-documented history (for example, medical record verification) in the 12 months prior to Screening Visit 1 of two or more moderate COPD exacerbations that were treated with systemic corticosteroids (intramuscular [IM], intravenous, or oral) with or without antibiotics or at least one severe COPD exacerbation requiring hospitalization.
* Participants must have a well-documented requirement for optimized standard of care background therapy that includes inhaled corticosteroids (ICS) plus 2 additional COPD medications (ICS-based triple therapy) for the 12 months prior to Screening Visit 1 and meets the following criteria: immediately prior to Screening Visit 1, minimum of 3 months of use of an 1) inhaled corticosteroid at a dose >=500 microgram (mcg) per day fluticasone propionate dose equivalent plus 2) Long acting beta2-agonist (LABA) and 3) Long acting muscarinic antagonist (LAMA) unless documentation of safety or intolerance issues related to LABA or LAMA. For participants who are not continually maintained on ICS plus LABA plus LAMA for the entire 12 months prior to Visit 1 use of the following is allowed (but not in the 3 months immediately prior to Visit 1); inhaled corticosteroid at a dose >=500 mcg per day fluticasone propionate dose equivalent plus inhaled LABA or inhaled LAMA and Phosphodiesterase-4-inhibitors, methylxanthines, or scheduled daily use of short acting beta2-agonist (SABA) and/or short acting muscarinic antagonist (SAMA).
* Current or former cigarette smokers with a history of cigarette smoking of >=10 pack-years at Screening (Visit 1) calculated as (number of pack years = [number of cigarettes per day/20] multiplied by number of years smoked [For example, 20 cigarettes per day for 10 years or 10 cigarettes per day for 20 years]).
* Contraceptive use for female participant should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: She is not a woman of childbearing potential (WOCBP) or she is a WOCBP and using a contraceptive method that is highly effective, with a failure rate of <1%, during the intervention period and for at least 16 weeks after the last dose of study intervention. The principal investigator (PI) should evaluate the effectiveness of the contraceptive method in relation to the first dose of study intervention.
* A WOCBP must have a negative highly sensitive pregnancy urine test within 24 hours before the first dose of study intervention. If a urine test cannot be confirmed as negative (For example, an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.
* Participants capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Participants must meet following randomization inclusion criteria at Visit 2 to be randomized and commence the study intervention period: a) Participants that do not have documented historical blood eosinophil count of ≥150 cells/μL prior to Screening Visit must meet this threshold based on the Screening Visit 1 assessment, b) Participants must have eosinophil count of ≥300 cells/μL from the hematology sample collected at Screening Visit 0, c) Compliance with completion of the e-diary defined as completion of all questions on 5 or more days out of the 7 days immediately preceding Visit 2.

Exclusion Criteria:

* Participants with a past history or concurrent diagnosis of asthma are excluded regardless of whether they have active or inactive disease.
* The Investigator must judge that COPD is the primary diagnosis accounting for the clinical manifestations of the lung disease. Participants with alpha1-antitrypsin deficiency as the underlying cause of COPD are excluded. Also, excluded are participants with active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, primary pulmonary hypertension, interstitial lung diseases or other active pulmonary diseases.
* Participants with pneumonia, COPD exacerbation, or lower respiratory tract infection within the 4 weeks prior to Screening Visit 1.
* Participants with lung volume reduction surgery within the 12 months prior to Screening Visit 1.
* Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Screening Visit 1. Participants who are in the maintenance phase of a pulmonary rehabilitation program are not excluded.
* Participants receiving treatment with oxygen more than 2 liter (L) per minute at rest over 24 hours. For participants receiving oxygen treatment, participants should demonstrate an oxyhemoglobin saturation greater than or equal to 89% while breathing supplemental oxygen.
* Participants with a QT interval, from the electrocardiogram (ECG) conducted at Screening Visit 1, corrected with Fridericia's formula (QTcF) >450 millisecond (msec) (or QTcF >480 msec in participants with bundle branch block). Fridericia's formula must be used to determine eligibility and discontinuation for an individual participant. Participants are excluded if an abnormal ECG finding from the 12-lead ECG conducted at Screening Visit 1 is considered to be clinically significant and would impact the participant's participation during the study, based on the evaluation of the Investigator.
* Participants with any of the following would be excluded: myocardial infarction or unstable angina in the 6 months prior to Screening Visit 1; unstable or life threatening cardiac arrhythmia requiring intervention in the 3 months prior to Screening Visit 1; New York Heart Association (NYHA) Class IV Heart failure.
* Participants with (historical or) current evidence of clinically significant, neurological, psychiatric, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities that are uncontrolled. Significant is defined as any disease that, in the opinion of the Investigator, would put the safety of the participant at risk through participation, or which could affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* Participants with other conditions that could lead to elevated eosinophils such as Hypereosinophilic syndromes including Eosinophilic Granulomatosis with Polyangiitis (EGPA), also known as Churg-Strauss Syndrome, or Eosinophilic Esophagitis.
* Participants with a known, pre-existing parasitic infestation within 6 months prior to Screening Visit 1.
* A current malignancy or previous history of cancer in remission for less than 12 months prior to Screening Visit 1 (participants that had localized carcinoma of the skin or cervix which was resected for cure will not be excluded).
* Participants with a known immunodeficiency (For example, human immunodeficiency virus [HIV]), other than that explained by the use of corticosteroids taken for COPD.
* Participants with cirrhosis or current unstable liver disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice. Stable non-cirrhotic chronic liver disease (including Gilbert's syndrome, asymptomatic gallstones, and chronic stable hepatitis B or C -e.g., presence of hepatitis B surface antigen [HbsAg] or positive hepatitis C antibody test result) is acceptable if the participant otherwise meets entry criteria.
* Participants who have received interventional product in previous mepolizumab studies are excluded.
* Participants who have received any monoclonal antibody within 5 half-lives of Screening Visit 1.
* Participants who have received an investigational drug within 30 days of Visit 1, or within 5 drug half-lives of the investigational drug, whichever is longer (this also includes investigational formulations of a marketed product).
* Participants who have received short term use of oral corticosteroids within 30 days of Visit 1.
* Participants with a known allergy or sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates participation in the study or intolerance to another monoclonal antibody or biologic including history of anaphylaxis to another biologic.
* Participants at risk of non-compliance, or unable to comply with the study procedures. Any infirmity, disability, or geographic location that would limit compliance for scheduled visits.
* Participants with conditions that will limit the validity of informed consent to participate in the study, for example, uncontrolled psychiatric disease or intellectual deficiency.
* Participants with a known or suspected history of alcohol or drug abuse within 2 years prior to Visit 1.
* Participant is an Investigator, sub-Investigator, study coordinator, employee of a participating Investigator or study site, or immediate family member of the aforementioned that is involved in this study.
* Participants with a current active COVID-19 infection, either laboratory confirmed or according to the investigator's medical judgement and who are known to be in contact with active COVID-19 positive individuals within the past 14 days.
* Participant will not be randomized if they meet any of the following randomization exclusion criteria at Visit 2: a) Participants who have pneumonia, exacerbation, lower respiratory infection during the Run-in period. b) Evidence of clinically significant abnormality in the hematological or biochemical screen at Visit 1, as judged by the Investigator. c) Participants who meet the following based on results from sample taken at Screening Visit 1: Alanine aminotransferase (ALT) >2x upper limit of normal (ULN), bilirubin >1.5 x ULN (isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%), cirrhosis or current unstable liver or biliary disease per Investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices, or persistent jaundice. d) Participants who are pregnant or breastfeeding. Participants should not be randomized if they plan to become pregnant during the time of study participation. e) Participants that had an active COVID-19 infection during the Run-in period, either laboratory confirmed or according to the investigator's medical judgment or known to be in contact with active COVID-19 positive individuals within the past 14 days. f) Participants with a QT interval, from the ECG conducted at Visit 2, corrected with Fridericia's formula (QTcF) >450 msec (or QTcF >480 msec in participants with bundle branch block).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 806 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (286):
- United States (88):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Dothan, Alabama
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Sheffield, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Gilbert, Arizona
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Conway, Arkansas
  - GSK Investigational Site, Alpine, California
  - GSK Investigational Site, Cerritos, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Boynton Beach, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Daytona Beach, Florida
  - GSK Investigational Site, Doral, Florida
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Homestead, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Miami Lakes, Florida
  - GSK Investigational Site, New Port Richey, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Pinellas Park, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Port Orange, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Adairsville, Georgia
  - GSK Investigational Site, Johns Creek, Georgia
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Woodstock, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Valparaiso, Indiana
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Natchitoches, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Lathrup Village, Michigan
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Toms River, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Gastonia, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Shelby, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Hilliard, Ohio
  - GSK Investigational Site, Kettering, Ohio
  - GSK Investigational Site, Norman, Oklahoma
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Altoona, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Clinton, South Carolina
  - GSK Investigational Site, Fort Mill, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Rock Hill, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Corsicana, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Lampasas, Texas
  - GSK Investigational Site, McAllen, Texas
  - GSK Investigational Site, McKinney, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Sherman, Texas
  - GSK Investigational Site, Webster, Texas
  - GSK Investigational Site, Rutland, Vermont
- Argentina (14):
  - GSK Investigational Site, Berazategui Buenos Aires
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad AutOnoma de Buenos Aire
  - GSK Investigational Site, Ciudad Autonoma de Bueno
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, La Plata
  - GSK Investigational Site, Lobos
  - GSK Investigational Site, Mar del Plata
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, Quilmes
  - GSK Investigational Site, Rosario
  - GSK Investigational Site, Rosario Provincia de Santa FE
  - GSK Investigational Site, San Miguel de Tucumán
  - GSK Investigational Site, San Rafael
- Australia (6):
  - GSK Investigational Site, Coffs Harbour, New South Wales
  - GSK Investigational Site, New Lambton, New South Wales
  - GSK Investigational Site, Sydney, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Kent Town, South Australia
  - GSK Investigational Site, Frankston, Victoria
- Belgium (3):
  - GSK Investigational Site, Jambes
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Yvoir
- Brazil (2):
  - GSK Investigational Site, Porto Alegre
  - GSK Investigational Site, São Paulo
- Canada (7):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Ajax, Ontario
  - GSK Investigational Site, Newmarket, Ontario
  - GSK Investigational Site, Sarnia, Ontario
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
- China (25):
  - GSK Investigational Site, Baotou
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Changchun
  - GSK Investigational Site, Changsha
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Hohehot
  - GSK Investigational Site, Jiaxing
  - GSK Investigational Site, Jinan
  - GSK Investigational Site, Nanchang
  - GSK Investigational Site, Nanjing
  - GSK Investigational Site, Nanning
  - GSK Investigational Site, Qingdao
  - GSK Investigational Site, Sanya
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Taiyuan
  - GSK Investigational Site, Taizhou
  - GSK Investigational Site, Ürümqi
  - GSK Investigational Site, Wuhan
  - GSK Investigational Site, Wuxi
  - GSK Investigational Site, Xiamen
  - GSK Investigational Site, Xining
  - GSK Investigational Site, Xinxiang
  - GSK Investigational Site, Zhuhai
  - GSK Investigational Site, Zigong
- Denmark (7):
  - GSK Investigational Site, Aalborg
  - GSK Investigational Site, Hvidovre
  - GSK Investigational Site, Kbenhavn N
  - GSK Investigational Site, Koebenhavn NV
  - GSK Investigational Site, Odense C
  - GSK Investigational Site, Roskilde
  - GSK Investigational Site, Vejle
- GSK Investigational Site, Tallinn, Estonia
- France (8):
  - GSK Investigational Site, Brest
  - GSK Investigational Site, Cholet
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Epagny Metz-Tessy
  - GSK Investigational Site, Le Mans
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Mulhouse
- Germany (18):
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Cottbus
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Fürstenwalde
  - GSK Investigational Site, Geesthacht
  - GSK Investigational Site, Gelsenkirchen
  - GSK Investigational Site, Halle
  - GSK Investigational Site, Immenhausen
  - GSK Investigational Site, Koblenz
  - GSK Investigational Site, Leipzig
  - GSK Investigational Site, Lübeck
  - GSK Investigational Site, Mainz
  - GSK Investigational Site, Neu-Isenburg
  - GSK Investigational Site, Peine
  - GSK Investigational Site, Rheine
  - GSK Investigational Site, Rodgau
  - GSK Investigational Site, Schleswig
  - GSK Investigational Site, Stuttgart
- Greece (5):
  - GSK Investigational Site, Alexandroupoli
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Ioannina
  - GSK Investigational Site, Rio Patras
  - GSK Investigational Site, Thessaloniki
- Hungary (9):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Gyula
  - GSK Investigational Site, Hajdúnánás
  - GSK Investigational Site, Hatvan
  - GSK Investigational Site, Pécs
  - GSK Investigational Site, Siófok
  - GSK Investigational Site, Törökbálint
  - GSK Investigational Site, Zalaegerszeg
- India (8):
  - GSK Investigational Site, Ahmedabad
  - GSK Investigational Site, Hyderabad
  - GSK Investigational Site, Jaipur
  - GSK Investigational Site, Kanpur
  - GSK Investigational Site, Lucknow
  - GSK Investigational Site, Nagpur
  - GSK Investigational Site, New Delhi
  - GSK Investigational Site, Puducherry
- Ireland (4):
  - GSK Investigational Site, Drogheda
  - GSK Investigational Site, Dublin
  - GSK Investigational Site, Galway
  - GSK Investigational Site, Limerick
- Israel (9):
  - GSK Investigational Site, Ashkelon
  - GSK Investigational Site, Beer-Yaakov
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Holon
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Ramat Gan
  - GSK Investigational Site, Rehovot
- Italy (5):
  - GSK Investigational Site, Bari
  - GSK Investigational Site, Ferrara
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Telese Terme BN
  - GSK Investigational Site, Verona
- Mexico (3):
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, Jalisco
  - GSK Investigational Site, Monterrey
- Netherlands (6):
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Heerlen
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, The Hague
  - GSK Investigational Site, Zutphen
- New Zealand (5):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Hamilton
  - GSK Investigational Site, Havelock North
  - GSK Investigational Site, Rotorua
  - GSK Investigational Site, Wellington
- Poland (18):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Częstochowa
  - GSK Investigational Site, Elblag
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Gdynia
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Kielce
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Ostrowiec Świętokrzyski
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Rzeszów
  - GSK Investigational Site, Sopot
  - GSK Investigational Site, Sosnowiec
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
  - GSK Investigational Site, Zamość
- South Korea (4):
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Jeonju
  - GSK Investigational Site, Seoul
- Spain (14):
  - GSK Investigational Site, Alzira
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Benalmádena
  - GSK Investigational Site, Cadiz
  - GSK Investigational Site, Cáceres
  - GSK Investigational Site, Galdakano
  - GSK Investigational Site, Granada
  - GSK Investigational Site, HebrOn
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marbella
  - GSK Investigational Site, Pozuelo de AlarcOn Madr
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Zaragoza
- Sweden (3):
  - GSK Investigational Site, Härnösand
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Uppsala
- Taiwan (2):
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
- United Kingdom (12):
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Cardiff
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Hardwick
  - GSK Investigational Site, Hexham
  - GSK Investigational Site, Lancashire
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Norwich
  - GSK Investigational Site, Reading
  - GSK Investigational Site, Wishaw

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Sciurba FC, Criner GJ, Christenson SA, Martinez FJ, Papi A, Roche N, Bourbeau J, Korn S, Bafadhel M, Han MK, Kolterer S, Miller K, Mouneimne D, Fletcher J, Mayer B, Min J, Pavord ID; MATINEE Study Investigators. Mepolizumab to Prevent Exacerbations of COPD with an Eosinophilic Phenotype. N Engl J Med. 2025 May 1;392(17):1710-1720. doi: 10.1056/NEJMoa2413181. PMID 40305712

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled 806 participants from multiple locations and regions worldwide.
Pre-assignment Details: Among the 806 participants, two were randomized in error and subsequently withdrawn from the study (one from the Mepolizumab 100 milligrams (mg) group and one from the Placebo group) without receiving any study intervention. The modified intention-to- treat (mITT) population consisted of 804 participants who were randomized and received at least one dose of the trial medication.
Period: Overall Study
Arm/Group | Mepolizumab 100 mg | Placebo
Started | 404 | 402
mITT Population | 403 | 401
Completed | 339 | 331
Not Completed | 65 | 71
Not completed — Death | 11 | 11
Not completed — Adverse Event | 4 | 5
Not completed — Lost to Follow-up | 3 | 5
Not completed — Physician Decision | 4 | 7
Not completed — Withdrawal by Subject | 40 | 35
Not completed — Lack of Efficacy | 2 | 7
Not completed — Randomized in error | 1 | 1

BASELINE CHARACTERISTICS:
Population: The analysis was performed on modified Intent-to-treat population (mITT) which included all randomized participants who received at least one dose of trial medication. Participants were analyzed by randomized treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mepolizumab 100 mg | Placebo | Total
Number analyzed (Participants) | 403 | 401 | 804
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 66.4 (8.10) | 66.0 (7.91) | 66.2 (8.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 126 | 253
  Male | 276 | 275 | 551
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — The 'All Other Races' category (Asian, American Indian or Alaska Native, Black or African American, and Mixed Race where 0<n<11) were combined into one category to maintain participant confidentiality and privacy.
  Participants
    White | 338 | 335 | 673
    All Other Races | 65 | 66 | 131

OUTCOME MEASURES:

1. Primary Outcome: Annualized Rate of Moderate or Severe Exacerbations
Description: Annualized rate of moderate or severe exacerbations were assessed. Moderate exacerbations are defined as clinically significant exacerbations that require treatment with oral or systemic corticosteroids and/or antibiotics. Severe exacerbations are defined per protocol as clinically significant exacerbations that require in-patient hospitalization (that is greater than or equal to [>=] 24 hours) or result in death.
Time Frame: Up to Week 104
Population: The analysis was performed on Modified Intent-to-Treat (mITT) population which included all randomized participants who received at least one dose of trial medication. Participants were analyzed by randomized treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Exacerbations per year
Arm/Group | Mepolizumab 100 mg | Placebo
Number analyzed (Participants) | 403 | 401
Exacerbations per year | 0.80 [0.70 to 0.91] | 1.01 [0.89 to 1.15]
Statistical Analysis 1: Comparison: Mepolizumab 100 mg vs Placebo; Analysis performed using a negative binomial model with covariates of treatment group, geographic region, number of moderate/severe exacerbations in previous year (less than or equal to [<=]2, 3, >=4 as ordinal), baseline percent (%) predicted Forced expiratory volume in one second (FEV1) and smoking status (current vs. former smoker), and with logarithm (time on- and off-treatment) as an offset variable; Test type: Superiority; p = 0.011, Negative binomial model; Rate ratio (Mepolizumab 100 mg/Placebo) = 0.79, 95% CI 2-sided [0.66 to 0.94]

2. Secondary Outcome: Time to First Moderate or Severe Exacerbation
Description: The time to first moderate or severe exacerbation was determined as the number of days from the date of first dose to the date of the first moderate or severe exacerbation. Kaplan-Meier estimate of the cumulative percentage of participants with a moderate or severe exacerbation within each treatment arm over time were produced.
Time Frame: At week 8,16, 24, 32, 40, 48, 52, 56, 64, 72, 80, 88, 96, 104
Population: The analysis was performed on mITT population which included all randomized participants who received at least one dose of trial medication. Participants were analyzed by randomized treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Mepolizumab 100 mg | Placebo
Number analyzed (Participants) | 403 | 401
Percentage of Participants
  At week 8 | 11.3 [8.5 to 14.8] | 15.1 [11.9 to 19.0]
  At week 16 | 21.6 [17.9 to 26.0] | 25.6 [21.6 to 30.2]
  At week 24 | 28.3 [24.2 to 33.1] | 35.4 [30.9 to 40.3]
  At week 32 | 33.6 [29.1 to 38.5] | 41.6 [36.9 to 46.7]
  At week 40 | 39.8 [35.1 to 44.8] | 47.1 [42.3 to 52.2]
  At week 48 | 44.9 [40.1 to 50.1] | 51.4 [46.6 to 56.5]
  At week 52 | 46.1 [41.2 to 51.2] | 53.4 [48.5 to 58.5]
  At week 56 | 46.7 [41.7 to 51.9] | 54.0 [49.0 to 59.2]
  At week 64 | 51.4 [45.8 to 57.2] | 58.9 [53.3 to 64.6]
  At week 72 | 55.9 [49.8 to 62.2] | 60.5 [54.7 to 66.4]
  At week 80 | 59.0 [52.6 to 65.5] | 62.3 [56.2 to 68.4]
  At week 88 | 60.6 [54.1 to 67.2] | 64.2 [57.9 to 70.5]
  At week 96 | 62.3 [55.6 to 69.0] | 67.2 [60.5 to 73.8]
  At week 104 | 64.5 [57.5 to 71.4] | 68.3 [61.4 to 74.9]
Statistical Analysis 1: Comparison: Mepolizumab 100 mg vs Placebo; Estimated from a Cox Proportional Hazards Model with covariates of treatment group, geographic region, number of moderate or severe exacerbations in previous year <=2, 3, >=4 as ordinal), baseline % predicted FEV1 and smoking status (current vs former); Test type: Superiority; p = 0.009, Cox Proportional Hazards Model; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.64 to 0.93]

3. Secondary Outcome: Percentage of COPD Assessment Test (CAT) Responders With >=2 Point Reduction From Baseline at Week 52
Description: The CAT is an 8-item questionnaire used to measure the health status of participants with COPD. Participants rated their experience on a 6-point scale, ranging from 0 (no impairment) to 5 (maximum impairment), with a scoring range of 0 (no impact)-40 (maximum impact). Higher scores indicate greater disease impact, and lower score indicates lesser disease impact. Participants were considered responders if they had a 2-point or more improvement (reduction) in CAT Score from baseline. Participants who withdrew from the study prior to Week 52 were included in the analysis as non-responders. The baseline value was the last measurement collected prior to the first dose of investigational product.
Time Frame: Baseline and Week 52
Population: The analysis was performed on mITT population which included all randomized participants who received at least one dose of trial medication. Participants were analyzed by randomized treatment. Only those participants with data available at the baseline were analyzed. Percentages were rounded-off to the nearest whole number.
Measure: Number; unit: Percentage of participants
Arm/Group | Mepolizumab 100 mg | Placebo
Number analyzed (Participants) | 391 | 394
Percentage of participants | 41 | 46
Statistical Analysis 1: Comparison: Mepolizumab 100 mg vs Placebo; A logistic regression model was used to compare the proportion of responders between the mepolizumab and placebo arms in the mITT and mITT2 populations. The model includes fixed categorical covariates (treatment group, smoking status, geographic region) and a fixed continuous covariate (baseline score); Test type: Superiority; p = 0.161, Regression, Logistic; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.60 to 1.09]

4. Secondary Outcome: Percentage of St. George's Respiratory Questionnaire for COPD (SGRQ) Total Score Responders With >=4 Point Reduction From Baseline at Week 52
Description: The St George's Respiratory Questionnaire for COPD (SGRQ-C) is a 40-item questionnaire. The total SGRQ score is calculated by summing up the weights of all positively answered items across the entire questionnaire, dividing by the total possible weight for all questionnaire items. The total score was expressed as a percentage of overall impairment, with 0 (best possible health status) and 100 (the worst possible health status). Higher scores indicated greater impairment of health, and lower scores indicate a lesser impairment on health. A participant was considered a responder if they had a 4-point or more improvement (reduction) in the SGRQ-C total score from baseline. Participants who withdrew from the study prior to Week 52 were included in the analysis as non- responders.
Time Frame: Baseline and Week 52
Population: The analysis was performed on mITT population which included all randomized participants who received at least one dose of trial medication. Participants were analyzed by randomized treatment. Only those participants with data available at the baseline were analyzed. Percentages were rounded off to the nearest whole number.
Measure: Number; unit: Percentage of participants
Arm/Group | Mepolizumab 100 mg | Placebo
Number analyzed (Participants) | 390 | 393
Percentage of participants | 50 | 46
Statistical Analysis 1: Comparison: Mepolizumab 100 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.291, Regression, Logistic; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.87 to 1.57]

5. Secondary Outcome: Percentage of Evaluating Respiratory Symptoms in COPD (E-RS: COPD) Responders With >=2 Point Reduction From Baseline
Description: The E-RS: COPD consists of 11 items from the 14 item Exacerbations of Chronic Pulmonary Disease Tool (EXACT) instrument (completed each evening using an eDiary). E-RS: COPD is intended to capture information related to the respiratory symptoms of COPD, that is, breathlessness, cough, sputum production, chest congestion, and chest tightness. The E-RS: COPD has a scoring range of 0 (no symptoms)-40 (most severe symptoms), higher scores indicate more severe symptoms. A participant is considered a responder if they have a 2-unit or more improvement (reduction) in their average E-RS: COPD total score during a 4-week period prior to Week 52 (Weeks 49-52) compared to baseline. The average of daily scores in 4-weekly intervals were calculated and data is presented for Weeks 49-52. Participants who withdrew from study prior to the start of the Weeks 49-52 time-period were included in the analysis as a non-responder.
Time Frame: Baseline and 4-weeks prior to Week 52
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Mepolizumab 100 mg | Placebo
Number analyzed (Participants) | 403 | 399
Percentage of participants | 31 | 34
Statistical Analysis 1: Comparison: Mepolizumab 100 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.209, Regression, Logistic; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.60 to 1.12]

6. Secondary Outcome: Annualized Rate of Exacerbations Requiring Emergency Department (ED) Visit and/or Hospitalization
Description: Annualized rate of exacerbations requiring ED visit or hospitalization were evaluated. This included moderate exacerbations which led to a visit to the ED and severe exacerbations, were defined as clinically significant exacerbations that require in-patient hospitalization (>= 24 hours) or result in death.
Time Frame: Up to Week 104
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Exacerbations per year
Arm/Group | Mepolizumab 100 mg | Placebo
Number analyzed (Participants) | 403 | 401
Exacerbations per year | 0.13 [0.10 to 0.18] | 0.20 [0.15 to 0.27]
Statistical Analysis 1: Comparison: Mepolizumab 100 mg vs Placebo; Analysis performed using a negative binomial model with covariates of treatment group, geographic region, number of moderate/severe exacerbations in previous year (<=2, 3, >=4 as ordinal), baseline % predicted FEV1 and smoking status (current vs. former smoker), and with logarithm (time on- and off-treatment) as an offset variable. Estimates based on weighting applied to each level of class variable determined from observed proportions; Test type: Superiority; p = 0.032, Negative binomial model; Rate ratio (Mepolizumab 100/Placebo) = 0.65, 95% CI 2-sided [0.43 to 0.96]

ADVERSE EVENTS:
Time Frame: Up to Week 104
Description: Data for All-Cause Mortality, Serious and Other (Non-Serious) Adverse Events were collected for the mITT population (all randomized participants, excluding those who were randomized in error). Safety population included all randomized participants who received at least one dose of trial medication.
Arm/Group | Mepolizumab 100 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 11/403 | 11/401
Serious Adverse Events (participants affected / at risk) | 101/403 | 115/401
Other Adverse Events (participants affected / at risk) | 195/403 | 182/401
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepolizumab 100 mg (N=403) | Placebo (N=401)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 3 (3)
Angina unstable (Cardiac disorders) | 2 (2) | 2 (2)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 4 (4) | 1 (1)
Cardiac failure (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (2) | 2 (2)
Coronary artery disease (Cardiac disorders) | 2 (2) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 3 (3)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 2 (2) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 2 (3)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bacterial pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 4 (4) | 6 (6)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (2)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 1 (1)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 5 (6)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 14 (16) | 17 (22)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 2 (3) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Scrotal abscess (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Stoma site abscess (Infections and infestations) | 0 (0) | 1 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumoconiosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Brain scan abnormal (Investigations) | 1 (1) | 0 (0)
Mycobacterium tuberculosis complex test negative (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tracheal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Parkinsonism (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 3 (3)
Device loosening (Product Issues) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 48 (74) | 56 (78)
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Angiokeratoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin plaque (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 1 (1)
Embolism arterial (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepolizumab 100 mg (N=403) | Placebo (N=401)
Diarrhoea (Gastrointestinal disorders) | 22 (23) | 12 (19)
COVID-19 (Infections and infestations) | 48 (52) | 47 (48)
Influenza (Infections and infestations) | 19 (24) | 18 (20)
Nasopharyngitis (Infections and infestations) | 41 (57) | 35 (46)
Pneumonia (Infections and infestations) | 18 (24) | 17 (20)
Upper respiratory tract infection (Infections and infestations) | 24 (40) | 20 (30)
Urinary tract infection (Infections and infestations) | 18 (20) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 (29) | 17 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 26 (46) | 23 (38)
Headache (Nervous system disorders) | 32 (62) | 28 (41)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 15 (17)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 (30) | 21 (38)
Hypertension (Vascular disorders) | 16 (16) | 26 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/09/NCT04133909/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-20): https://cdn.clinicaltrials.gov/large-docs/09/NCT04133909/SAP_001.pdf